CLINICAL TRIAL: NCT05792956
Title: The Effect of Mobile Application and Bladder Training on Quality of Life and Sexual Satisfaction in Women With Overactive Bladder
Brief Title: Mobile Application and Bladder Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Nurdan Demirci, Prof, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Mu_olmezyalazi
Record Dates: First submitted 2023-03-13; First posted 2023-03-31 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Overactive Bladder Syndrome
Keywords: Overactive bladder; Mobile application; Quality of life; Sexual satisfaction
MeSH Terms: conditions — Urinary Bladder, Overactive; Orgasm

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Application group (Experimental): Women with OAB in this group will be informed about mobile application usage. The group using the mobile application will add the times they have consumed fluid and urine leakage to the bladder diary section of the mobile application. During the day, the application will remind participants to consume fluids and urinate. There will also be a question and answer section in the mobile application. Women will be able to direct their questions about OAB to the researcher. After the first meeting, the scales sent through the mobile application will be applied in the 3rd and 6th months.
  Interventions: Behavioral: Using mobile app
- Control group (No Intervention): To the control group, the routine protocol in the clinic (Bladder training is given by the nurses after the women apply. They come to deliver the bladder diary given after the bladder training in the 3rd and 6th months. According to the results of the bladder diary, the nurses provide counseling for the problems detected regarding the symptoms they experience). After the first interview, they will be asked to fill in the required scales one day in the 3rd and 6th months.

INTERVENTIONS:
Behavioral: Using mobile app — Women with OAB in this group will be informed about mobile application usage. The group using the mobile application will add the times they have consumed fluid and urine leakage to the bladder diary section of the mobile application. During the day, the application will remind participants to consume fluids and urinate. There will also be a question and answer section in the mobile application. Women will be able to direct their questions about OAB to the researcher. After the first meeting, the scales sent through the mobile application will be applied in the 3rd and 6th months.
  Arms: Mobile Application group

SUMMARY:
The International Continence Society described overactive bladder as urine urgency, frequently accompanied by frequency and nocturia, with or without urgency incontinence, when there is no evident pathology, such as a urinary tract infection. According to studies in the literature, women who have overactive bladders experience negative effects on their sexual satisfaction and quality of life. According to a study by Juliato et al. (2017), women with more severe urinary symptoms experienced higher degrees of arousal, lubrication, orgasm, and discomfort. According to Chuang et al. (2017) study, women's sexual pleasure and quality of life declined as urinary symptom intensity increased. It is believed that women's quality of life and levels of sexual satisfaction may be positively impacted by the training provided to lessen their symptoms, their follow-up, and their continuity. Additionally, it is anticipated that by encouraging better treatment compliance among women with OAB, hospital expenses will drop, which will benefit the national economy. In order to ascertain the impact of bladder training delivered via mobile application on quality of life and levels of sexual satisfaction in women with overactive bladder, this study was designed.

Between February 2023 and June 2024, this randomized controlled experimental design study will be conducted in the urogynecology clinic of a university hospital on Istanbul's Anatolian side. The sample size was determined via G-Power power analysis, and the groups were chosen using basic randomization. There will be 100 women studied, 50 in the study group (WG) and 50 in the control group (KG), all of whom have been diagnosed with overactive bladder. Through the smartphone application, WG women will receive bladder training, as well as follow-up care. Data will be gathered using the Quality of Life Scale, Sexual Satisfaction Scale, Mobile Application Usage Scales (only mobile application group), and Collection Form, Follow-Up Form. In the third and sixth months, new data will be collected on the Quality of Life Scale, Sexual Satisfaction Scale, and Mobile Application Usage Scales (just for the Mobile Application Group). There will be a data analysis.

DETAILED DESCRIPTION:
According to the International Continence Society (ICS), overactive bladder (OAB), usually accompanied by increased urination during the day or nocturia, is defined as a serious symptom of urinary incontinence that occurs without urinary tract infection or other diagnosable disease. The prevalence of OAB ranges from 12-22% in Europe and 16-17% in the USA. According to a comprehensive study conducted in Turkey in 2014, the prevalence of urgent urinary incontinence, which is mostly seen in individuals diagnosed with OAB, was reported as 29.3%. Although the prevalence of OAB is similar in men and women, various symptoms of OAB can be seen more in women due to anatomical and physiological differences in the lower urinary tract. OAB affects an individual's daily life, including work, social interactions, sleep patterns, and sexual functions. In studies, it has been reported that women diagnosed with OAB tend to increase in sleep disorders, affect normal social activities, decrease sexuality and quality of life, and impair self-esteem. In a study by Juliato et al. (2017), it was reported that arousal, lubrication, orgasm and pain levels increased in women with high urinary symptom severity (according to the ICIQ-OAB score). In the study of Chuang et al. (2019), it was determined that increased urinary symptom severity in women decreased sexual satisfaction and quality of life levels. It is of great importance to choose an effective and treatment method for women diagnosed with OAB. There are 3 types of treatment methods to alleviate OAB symptoms: Pharmacological (second-line treatment), non-pharmacological (first and third-line treatments), and surgical intervention. The American Urological Association (AUA) and Urogynecology Society, Female Pelvic Medicine and Pelvic Reconstruction (SUFU) guidelines recommend that OAB be treated step by step, starting with the least invasive treatment. Due to the concern about the side effects of the given drug and the complications of invasive procedures, non-pharmacological interventions are an important part of the treatment of OAB. Antimuscarinics such as solifenacin are used after unsuccessful conservative and behavioral treatments. However, due to the high cost and the presence of side effects (such as dry mouth, headache, constipation and visual irregularity), women's compliance with these drugs decreases and consequently limits their use. However, minimally invasive procedures have risks and complications. In addition, the healing process is supported by non-pharmacological methods after minimally invasive treatment. According to the results of the studies, it was reported that 31-40% of women were supported by non-pharmacological treatment method after minimally invasive intervention. Among the non-pharmacological treatment methods for OAB, bladder training is thought to be the most effective. It has been reported that the training, follow-up and continuity of women to reduce their symptoms can increase their quality of life and sexual satisfaction levels. It is thought that due to the cost of the treatments, the problems of compliance with the treatment process, the decrease in sustainability and the limited accessibility of healthcare professionals, bladder training can be used to increase the compliance and sustainability of women to the treatment process by using different methods. It is thought that it can be used to follow and maintain the training given with the user interface with mobile applications. Therefore, it is important in terms of patient satisfaction and sustainability as well as reducing the cost of treatment. The mobile application the investigators will develop will be an educational tool in the digital environment that allows nurses to communicate with patients, follow the treatment process and enable women to be active in process management. It is aimed to ensure continuity by optimizing the individualized care and well-being of women in line with the results, and accordingly, to minimize the complications that may occur as a result of other treatment methods. Therefore, the effect of the mobile application-based training and notifications the investigators will develop on the quality of life and sexual satisfaction levels in women will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers aged 18 and over,
* Diagnosed with OAB,
* Being literate and having no communication problems,
* Does not have a mental problem that requires treatment,
* Not mentally handicapped, hearing impaired, visually impaired, language and speech impaired,
* Not diagnosed with a psychiatric disorder,
* Able to use a smart phone,
* Women who can speak Turkish will be included in the study.

Exclusion Criteria:

* Emergency operation during the research,
* Not filling in the forms submitted to evaluate the symptoms,
* Being in the mobile application group and not using the application,
* Those who do not agree to participate in the research, Women who became pregnant during the study will not be included.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Number of Overactive Bladder have women | 6 month
  In the study, R v3.6.1 program was used for Power analysis, alpha error was 5%, beta error was 20%, it was predicted that there would be a difference between the variables as a result of the study process, and a minimum of 100 (50 mobile application groups, 50 control groups) samples would be sufficient.

SECONDARY OUTCOMES:
Evaluation of symptoms | First, 3rd and 6th months
  Symptoms will be evaluated at 3 and 6 months after the first interview
Mobile application scales evaluation | 3rd and 6th months
  The group using the mobile application will evaluate the effectiveness of the mobile application with the scales* for evaluating the mobile application in the 3rd and 6th months.
  * The Mobile Application Usability Scale is a scale consisting of 10 factors, each of which has 4 items, and a total of 40 items. The scale is a likert-type scale scored from 1 to 7. As the total score increases, the level of mobile application usability also increases.
  * Willingness to Use Mobile Application Scale, Single factor, 6-item scale, from 1 to 7 is a likert-type scale. As the total score increases, the level of willingness to use mobile applications also increases.
  * Mobile Application Loyalty Scale, Single factor, 5-item scale, from 1 to 7. As the total score increases, the loyalty level of using mobile applications also increases.
Evaluation of quality of life | First, 3rd and 6th months
  The first interview of both groups will evaluate their quality of life with the quality of life scale* in the 3rd and 6th months.
  *International Consultation on Incontinence Questionnaire-lower urinary tract symptoms-quality of life (ICIQ-LUTSqol) is an ideal research tool as it explores in detail the impact on patients' lives of urinary incontinence and can be used as an outcome measure to assess impact of different treatment modalities.19-76 overall score with greater values indicating increased impact on quality of life Bother scales are not incorporated in the overall score but indicate impact of individual symptoms for the patient.
• New Sexual Satisfaction Scale | First, 3rd and 6th months
  Both groups will evaluate their sexual satisfaction levels with the sexual satisfaction scale* at the first interview, at the 3rd and 6th months.
  *The scale was developed to measure sexual satisfaction in the clinical and field studies and has a 5-Likert structure. Scoring of the scale is calculated by summing the items points. The minimum and maximum scores that can be received from the scale are 20 and 100 points, respectively. High scores from the scale indicate high sexual satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Rüveyda ölmez yalazı, PhDc, Principal Investigator — Marmara University; Nurdan Demirci, Prof, Study Director — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No